CLINICAL TRIAL: NCT03468062
Title: The Effect of Preoperative Intravenous Dexmedetomidine on Postoperative Quality of Recovery: Randomized Study
Brief Title: The Effect of Dexmedetomidine on Postoperative Quality of Recovery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kyungmi Kim (Other)
Responsible Party: Sponsor-Investigator, Kyungmi Kim, Assistant Professor, Gachon University Gil Medical Center
Organization: Gachon University Gil Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GAIRB2018-071
Record Dates: First submitted 2018-03-11; First posted 2018-03-16 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: The Effect of Dexmedetomidine on Postoperative Quality of Recovery
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): 0.5 mg/kg of dexmedetomidine (Precedex; Hospira, Lake Forest, IL) is mixed in normal saline 100mL and administered for 5 minutes after anesthetic induction.
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Only normal saline 100mL is administered for 5 minutes after anesthetic induction.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Patients assigned in Dexmedetomidine or Placebo group are given Dexmedetomidine or normal saline after induction of anesthesia.
  Other Names: Placebo

SUMMARY:
Dexmedetomidine is a selective a2-agonist and a sedative with anti-inflammatory,analgesic, and antiemetic effects, and its use for procedural sedation during endoscopy or ablation for atrial fibrillation has been increasing. It is also used for sedation in the intensive care unit. Recently, it was reported that dexmedetomidine is often used as an adjuvant for general anesthesia. Sympatholysis of dexmedetomidine can attenuate the increased sympathetic tone after surgery and result in antistress effects. In addition, opioid-sparing and analgesic effects are promoted by the perioperative administration of dexmedetomidine. Although it has been reported that the perioperative administration of dexmedetomidine improves quality of recovery after spinal and ENT surgeries, the outcomes for patients who undergo laparoscopic cholecystectomy remain poorly investigated.

The aims of this study were to evaluate the effects of preoperative dexmedetomidine administration on quality of recovery by using the QoR-40 questionnaire in patients who undergo laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* The patients who undergo elective cholecystectomy
* Adults (20~75 years old)
* an American Society of Anesthesiologists physical status of I or II

Exclusion Criteria:

* The patients do not provide written informed consent
* The patients have had allergic response to dexmedetomidine.
* The patients have mood disorder or anxiety disorder.
* The patients are not able to express their emotions.
* The pregnant women

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery questionnaire | postoperative first day
  The Quality of Recovery questionnaire (QoR-40) is a tool used to assess the quality of recovery after surgery through questions pertaining to 40 items related to 5 domains. It has been validated as a global and reliable measurement tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Gil Medical Center, Gachon University College of Medicine, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi JJ, Kim K, Park HY, Chang YJ, Lee KC, Kim KY, Kwak HJ. CONSORT the effect of a bolus dose of dexmedetomidine on postoperative pain, agitation, and quality of recovery after laparoscopic cholecystectomy. Medicine (Baltimore). 2021 Jan 22;100(3):e24353. doi: 10.1097/MD.0000000000024353. PMID 33546069